CLINICAL TRIAL: NCT06001463
Title: CSMed Wound Dressing on Radiation Dermatitis Clinical Trial
Brief Title: Clinical Trial of CSMed Wound Dressing for Radiation Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Yueh-Chun Lee, Radiation Oncology Attending Physician, Chung Shan Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1 20015
Record Dates: First submitted 2023-02-21; First posted 2023-08-21 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- reduce the severity, and enhance healing of radiation dermatitis (Experimental): The patient received part of the breast/neck skin CSMed® dressing or clinical routine skin care.
  Interventions: Drug: CSMed Dressing

INTERVENTIONS:
Drug: CSMed Dressing — Half of the irradiated area was covered with CSMed® and the other half was under routine treatment. An irradiated area of 11cm*14cm with best fit or easy accessibility was chosen for CSMed® dressing application. The area without dressing was treated with routine skin care in each patient.

SUMMARY:
Investigate the effects of CSMed® for preventing and managing radiation dermatitis in patients with Breast cancer and Head-Neck cancer receiving radiotherapy (≥50 Gy).

DETAILED DESCRIPTION:
A prospective study was conducted at the University Hospital Medical Center. The patient received part of the breast/neck skin CSMed® dressing or clinical routine skin care. Record the difference between the part of the skin with dressing and undressed skin for each patient. The severity of acute radiation dermatitis was graded using the RTOG clinical scoring standard. From the beginning of the treatment to 4 weeks after the end of the treatment, skin pain, itching, local fever and tightness, as well as skin healing time were collected every week.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving radiation therapy (including undamaged skin and RTOG grade 1 dermatitis).
* Patients who voluntarily agree to participate in the trial and sign the subject's consent form.

Exclusion Criteria:

* Patients with dermatitis and burns not caused by radiation therapy.
* Involuntary patients without signed consent.
* Those who are allergic to the ingredients in this product.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Severity of acute radiation dermatitis | 4 weeks
  The severity of radiation dermatitis can be assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE). Grade 1 to 5.
  NCI CTCAE grade 1 - Faint erythema with dry desquamation. NCI CTCAE grade 2 - Moderate dermatitis is characterized by moderate to brisk erythema and patchy, moist desquamation mostly confined to skin folds and creases.
  NCI CTCAE grade 3 - There is confluent, moist desquamation in locations other than skin folds.
  NCI CTCAE grade 4 - This is characterized by skin necrosis or ulceration of full-thickness dermis.
  NCI CTCAE grade 5 - Death due to dermatitis alone is a very rare event.
  Radiologists performed radiation therapy according to the needs of clinical diseases. Evaluate and record the case after radiotherapy at 4 weeks, and end the research record.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No